CLINICAL TRIAL: NCT02368002
Title: Evaluating Options for Non-Responders: A SMART Approach to Enhancing Weight Loss
Brief Title: BestFIT: a Personalized Weight Loss Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: Drexel University (Other); University of Michigan (Other); University of Minnesota (Other); University of Washington (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1R01CA188892-01 (NIH); 1R01CA188892-01 (NIH)
Record Dates: First submitted 2015-02-06; First posted 2015-02-20 (Estimated); Results first posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2019-07

CONDITIONS: Obesity
Keywords: obesity; diet, reducing
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Behavioral weight loss therapy (Experimental): Emphasizes 1) identifying behaviors in need of change, 2) setting goals for change, 3) monitoring progress, 4) modifying environmental cues to facilitate change, and 5) modifying consequences to motivate change.
  Interventions: Behavioral: Behavioral weight loss therapy
- Portion-controlled meals (Experimental): Fifty percent of participants who have not lost the expected amount of weight will be re-randomized to receive portion-controlled meals in addition to standard behavioral weight loss therapy.
  Interventions: Behavioral: Portion-controlled meals
- Acceptance-based treatment (Experimental): Fifty percent of participants who have not lost the expected amount of weight will be re-randomized to receive an enhanced version of behavioral weight loss therapy teaching acceptance-based behavioral skills.
  Interventions: Behavioral: Acceptance-based treatment

INTERVENTIONS:
Behavioral: Behavioral weight loss therapy — All participants start with behavioral weight loss therapy which consists of 20 weekly meetings wtih a weight loss coach. Session components will include weekly weigh-in, discussion of progress and challenges and discussion of scheduled session topic. Dietary goals and physical activity goals are set. After their first session, participants are randomized to have their weight assessed at either their 3rd session or their 7th session. Both the participant and their coach are blinded to the randomization. If the participant has lost the expected amount of weight, they continue with behavioral weight loss therapy for the full 20 session.
  Arms: Behavioral weight loss therapy
Behavioral: Portion-controlled meals — Participants continue with behavioral weight loss therapy, but this is augmented with portion-controlled meals (PCM). Adherence to energy intake goals is facilitated by consuming pre-prepared meals specifically designed to meet caloric intake guidelines. PCMs reduce individuals' motivationally- and self-regulatory-dependent planning and decision making around eating. PCMs also serve as a "teaching tool" regarding the amount and type of food people should eat in order to produce weight loss.
  Arms: Portion-controlled meals
Behavioral: Acceptance-based treatment — Switching the therapeutic approach to an enhanced behavioral weight loss therapy teaching acceptance-based behavioral skills theoretically addresses the root problem of many weight loss challenges and boosts long-term capacity for self-regulation. Acceptance based strategies are designed to help participants identify and internalize values and lasting commitment to behavior consistent with these values. The strategies focus on increasing people's ability to forgo more pleasurable options (e.g., hedonic pleasure of food) in favor of behavior that is distinctly less pleasurable or even aversive (remaining hungry, anxious, bored). The inability to tolerate such distress is directly associated with failure of self-regulation.
  Arms: Acceptance-based treatment

SUMMARY:
The purpose of this study is to learn how to personalize weight loss programs. In this research we will study:

1. Whether a weight loss counselor should decide if the traditional weight loss therapy is working either after 3 or 7 weekly sessions of therapy and
2. For those who haven't lost the expected amount of weight, whether it is more effective to add packaged meals to the traditional weight loss therapy or to change to an enhanced version of behavioral weight loss therapy.

DETAILED DESCRIPTION:
The US Preventive Services Task Force recommends referral to behavioral weight loss programs to help obese adults achieve a clinically meaningful weight loss of 8-10% of starting body weight. However, approximately half of participants are unable to achieve this goal. Despite this, a"one size fits all" approach is the norm, a major drawback because those who do not respond can in fact be detected early. This gap in weight loss intervention science calls for an adaptive intervention approach that could provide the "right treatment at the right time for the right person". Adaptive interventions individualize treatment through empirically-supported decision rules advising when and how treatments should unfold over time to maximize effectiveness. Sequential Multiple Assignment Randomized Trials (SMART), developed explicitly to build the best adaptive interventions, use experimental design principles to develop these decision rules. The investigators will use a SMART to systematically evaluate therapeutic approach and timing differences for intervening with those who do not respond to a behavioral weight loss program. Self-regulation challenges have been identified as a major adherence barrier. Two attractive options to address self-regulation difficulties are: 1) supplementing behavioral treatment with Meal Replacements (MR) which decreases the need for self-regulation; and 2) switching therapeutic approaches by using an enhanced version of behavioral weight loss therapy that teaches acceptance based behavioral skills which boost capacity for self-regulation. Additionally, two time points for intervening with non-responders will be evaluated: 1) 3 weeks, based on current weight loss trial evidence; and 2) 7 weeks, based on average time used in the existing stepped care literature. Adults (n=500) will be recruited and will receive individual behavioral weight loss treatment (BWL). Participants will be randomized to either: 1) treatment response assessment at 3 weeks or 2) treatment response assessment at 7 weeks. Subjects who have lost the expected amount of weight at their assessment point, will continue with traditional behavioral weight loss therapy. For those who have not lost the expected amount of weight, we will re-randomize them to either meal replacements in addition to the traditional weight loss therapy or to the enhanced version of behavioral weight loss therapy.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 21 - 70
* BMI between 30 - 45 kg/m2
* Able to walk 2 blocks without stopping
* Able to attend measurement and intervention activities in the Twin Cities area in person for 18 months

Exclusion Criteria:

* Self-reported pregnancy or breastfeeding baby in last 6 months or planning a pregnancy in the next 18 months
* History of bariatric surgery
* Current or previous diagnosis of anorexia nervosa or bulimia nervosa
* Food allergies, intolerances

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy E Sherwood, PhD, Principal Investigator — University of Minnesota; A. Lauren Crain, PhD, Principal Investigator — HealthPartners Institute
Locations (1):
- HealthPartners Institute, Bloomington, Minnesota, United States

REFERENCES:
- [Background] Carels RA, Darby L, Cacciapaglia HM, Douglass OM, Harper J, Kaplar ME, Konrad K, Rydin S, Tonkin K. Applying a stepped-care approach to the treatment of obesity. J Psychosom Res. 2005 Dec;59(6):375-83. doi: 10.1016/j.jpsychores.2005.06.060. PMID 16310019
- [Background] Lei H, Nahum-Shani I, Lynch K, Oslin D, Murphy SA. A "SMART" design for building individualized treatment sequences. Annu Rev Clin Psychol. 2012;8:21-48. doi: 10.1146/annurev-clinpsy-032511-143152. Epub 2011 Dec 12. PMID 22224838
- [Background] Collins LM, Murphy SA, Strecher V. The multiphase optimization strategy (MOST) and the sequential multiple assignment randomized trial (SMART): new methods for more potent eHealth interventions. Am J Prev Med. 2007 May;32(5 Suppl):S112-8. doi: 10.1016/j.amepre.2007.01.022. PMID 17466815
- [Background] Butryn ML, Webb V, Wadden TA. Behavioral treatment of obesity. Psychiatr Clin North Am. 2011 Dec;34(4):841-59. doi: 10.1016/j.psc.2011.08.006. PMID 22098808
- [Background] Rock CL, Flatt SW, Sherwood NE, Karanja N, Pakiz B, Thomson CA. Effect of a free prepared meal and incentivized weight loss program on weight loss and weight loss maintenance in obese and overweight women: a randomized controlled trial. JAMA. 2010 Oct 27;304(16):1803-10. doi: 10.1001/jama.2010.1503. Epub 2010 Oct 9. PMID 20935338
- [Background] Heymsfield SB, van Mierlo CA, van der Knaap HC, Heo M, Frier HI. Weight management using a meal replacement strategy: meta and pooling analysis from six studies. Int J Obes Relat Metab Disord. 2003 May;27(5):537-49. doi: 10.1038/sj.ijo.0802258. PMID 12704397
- [Background] Forman EM, Hoffman KL, McGrath KB, Herbert JD, Brandsma LL, Lowe MR. A comparison of acceptance- and control-based strategies for coping with food cravings: an analog study. Behav Res Ther. 2007 Oct;45(10):2372-86. doi: 10.1016/j.brat.2007.04.004. Epub 2007 Apr 18. PMID 17544361
- [Background] Sherwood NE, Butryn ML, Forman EM, Almirall D, Seburg EM, Lauren Crain A, Kunin-Batson AS, Hayes MG, Levy RL, Jeffery RW. The BestFIT trial: A SMART approach to developing individualized weight loss treatments. Contemp Clin Trials. 2016 Mar;47:209-16. doi: 10.1016/j.cct.2016.01.011. Epub 2016 Jan 26. PMID 26825020
- [Derived] Emery Tavernier RL, Mason SM, Levy RL, Seburg EM, Sherwood NE. Association of childhood abuse with behavioral weight-loss outcomes: Examining the mediating effect of binge eating severity. Obesity (Silver Spring). 2022 Jan;30(1):96-105. doi: 10.1002/oby.23320. PMID 34932887
- [Derived] Sherwood NE, Crain AL, Seburg EM, Butryn ML, Forman EM, Crane MM, Levy RL, Kunin-Batson AS, Jeffery RW. BestFIT Sequential Multiple Assignment Randomized Trial Results: A SMART Approach to Developing Individualized Weight Loss Treatment Sequences. Ann Behav Med. 2022 Mar 1;56(3):291-304. doi: 10.1093/abm/kaab061. PMID 34415011
- [Derived] Crane MM, Seburg EM, Levy RL, Jeffery RW, Sherwood NE. Using targeting to recruit men and women of color into a behavioral weight loss trial. Trials. 2020 Jun 16;21(1):537. doi: 10.1186/s13063-020-04500-1. PMID 32546253

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 26 participants were lost to follow-up or quit after the initial randomization to the 3 or 7 week treatment response assessment and prior to the treatment response assessment. These participants are included in the session 3 and session 7 treatment response assessment & no-randomization groups.
Groups:
- Session 3 Treatment Response Assessment: Participants randomized to treatment response assessment at session 3. All participants start with standard behavioral weight loss treatment, and treatment response assessment occurs at session 3. If participants lost the expected amount of weight, no re-randomization occurs and participants continue with standard behavioral weight loss treatment. If participants did not lose the expected amount of weight, re-randomization to PCM or ABT occurs.
- Session 3 Treatment Response Assessment & ABT: Participants randomized to treatment response assessment at session 3 and re-randomized to acceptance-based treatment (ABT). Participants started with standard behavioral weight loss treatment. Participants did not lose the expected amount of weight at the session 3 treatment response assessment and were re-randomized to switch to ABT.
- Session 3 Treatment Response Assessment & PCM: Participants randomized to treatment response assessment at session 3 and re-randomized to portion controlled meals (PCM). Participants started with standard behavioral weight loss treatment. Participants did not lose the expected amount of weight at the session 3 treatment response assessment and were re-randomized to behavioral weight loss therapy augmented with PCM.
- Session 7 Treatment Response Assessment: Participants randomized to treatment response assessment at session 7. All participants start with standard behavioral weight loss treatment, and treatment response assessment occurs at session 7. If participants lost the expected amount of weight, no re-randomization occurs and participants continue with standard behavioral weight loss treatment. If participants did not lose the expected amount of weight, re-randomization to PCM or ABT occurs.
- Session 7 Treatment Response Assessment & ABT: Participants randomized to treatment response assessment at session 7 and re-randomized to acceptance-based treatment (ABT). Participants started with standard behavioral weight loss treatment. Participants did not lose the expected amount of weight at the session 7 treatment response assessment and were re-randomized to switch to ABT.
- Session 7 Treatment Response Assessment & PCM: Participants randomized to treatment response assessment at session 7 and re-randomized to portion controlled meals (PCM). Participants started with standard behavioral weight loss treatment. Participants did not lose the expected amount of weight at the session 7 treatment response assessment and were re-randomized to behavioral weight loss therapy augmented with PCM.
Period: Stage 1 Intervention (Up to 20 Weeks)
Arm/Group | Session 3 Treatment Response Assessment | Session 3 Treatment Response Assessment & ABT | Session 3 Treatment Response Assessment & PCM | Session 7 Treatment Response Assessment | Session 7 Treatment Response Assessment & ABT | Session 7 Treatment Response Assessment & PCM
Started | 233 | 0 | 0 | 235 | 0 | 0
Completed | 228 | 0 | 0 | 214 | 0 | 0
Not Completed | 5 | 0 | 0 | 21 | 0 | 0
Period: Stage 2 Intervention (Up to 17 Weeks)
Arm/Group | Session 3 Treatment Response Assessment | Session 3 Treatment Response Assessment & ABT | Session 3 Treatment Response Assessment & PCM | Session 7 Treatment Response Assessment | Session 7 Treatment Response Assessment & ABT | Session 7 Treatment Response Assessment & PCM
Started | 88 | 70 | 70 | 0 | 0 | 0
Completed | 86 | 60 | 64 | 0 | 0 | 0
Not Completed | 2 | 10 | 6 | 0 | 0 | 0
Period: Stage 2 Intervention (Up to 13 Weeks)
Arm/Group | Session 3 Treatment Response Assessment | Session 3 Treatment Response Assessment & ABT | Session 3 Treatment Response Assessment & PCM | Session 7 Treatment Response Assessment | Session 7 Treatment Response Assessment & ABT | Session 7 Treatment Response Assessment & PCM
Started | 0 | 0 | 0 | 95 | 57 | 62
Completed | 0 | 0 | 0 | 94 | 53 | 59
Not Completed | 0 | 0 | 0 | 1 | 4 | 3

BASELINE CHARACTERISTICS:
Population: Participants who were re-randomized to a second line treatment (PCM or ABT) are represented more than once in the Total Arm/Group. They are included in either the Week 3 or Week 7 treatment response assessment group and the Portion controlled meals or Acceptance-based treatment group.
Groups:
- Week 3 Treatment Response Assessment: Participants randomized to have their weight assessed at their 3rd session. If the participant has lost the expected amount of weight, they continue with standard behavioral weight loss treatment for the full 20 sessions. If they have not lost the expected amount of weight, they are re-randomized to portion controlled meals or acceptance-based treatment.
- Week 7 Treatment Response Assessment: Participants randomized to have their weight assessed at their 7th session. If the participant has lost the expected amount of weight, they continue with standard behavioral weight loss treatment for the full 20 sessions. If they have not lost the expected amount of weight, they are re-randomized to portion controlled meals or acceptance-based treatment.
- Portion Controlled Meals: Portion controlled meals: Participants assessed at the 3rd or 7th session who did not lose the expected amount of weight and were re-randomized to continue with behavioral weight loss therapy that is augmented with portion controlled meals (PCM).
- Acceptance-based Treatment: Acceptance-based treatment: Participants assessed at the 3rd or 7th session who did not lose the expected amount of weight and were re-randomized to switching the therapeutic approach to an acceptance-based treatment.
- Total: Total of all reporting groups
Arm/Group | Week 3 Treatment Response Assessment | Week 7 Treatment Response Assessment | Portion Controlled Meals | Acceptance-based Treatment | Total
Number analyzed (Participants) | 233 | 235 | 132 | 127 | 727
Age, Categorical [Count of Participants; unit: Participants] — Population: We report data for two periods: "Stage 1 Randomization" (initial randomization to Week 3 or Week 7 Treatment Response Assessment) and "Stage 2 Re-Randomization" (re-randomization of sub-optimal responders to Portion controlled meals or Acceptance-based treatment).
  Participants
    Stage 1 Randomization: number analyzed (Participants) | 233 | 235 | 0 | 0 | 468
    Stage 1 Randomization: <=18 years | 0 | 0 |  |  | 0
    Stage 1 Randomization: Between 18 and 65 years | 224 | 225 |  |  | 449
    Stage 1 Randomization: >=65 years | 9 | 10 |  |  | 19
    Stage 2 Re-Randomization: number analyzed (Participants) | 0 | 0 | 132 | 127 | 259
    Stage 2 Re-Randomization: <=18 years |  |  | 0 | 0 | 0
    Stage 2 Re-Randomization: Between 18 and 65 years |  |  | 125 | 125 | 250
    Stage 2 Re-Randomization: >=65 years |  |  | 7 | 2 | 9
Sex: Female, Male [Count of Participants; unit: Participants] — Population: We report data for two periods: "Stage 1 Randomization" (initial randomization to Week 3 or Week 7 Treatment Response Assessment) and "Stage 2 Re-Randomization" (re-randomization of sub-optimal responders to Portion controlled meals or Acceptance-based treatment).
  Participants
    Stage 1 Randomization: number analyzed (Participants) | 233 | 235 | 0 | 0 | 468
    Stage 1 Randomization: Female | 179 | 178 |  |  | 357
    Stage 1 Randomization: Male | 54 | 57 |  |  | 111
    Stage 2 Re-Randomization: number analyzed (Participants) | 0 | 0 | 132 | 127 | 259
    Stage 2 Re-Randomization: Female |  |  | 111 | 111 | 222
    Stage 2 Re-Randomization: Male |  |  | 21 | 16 | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Participants who were re-randomized to a second line treatment (PCM or ABT) are represented more than once in the Total Arm/Group. They are included in either the Week 3 or Week 7 treatment response assessment group and the Portion controlled meals or Acceptance-based treatment group.
  Participants
    Stage 1 Randomization: number analyzed (Participants) | 233 | 235 | 0 | 0 | 468
    Stage 1 Randomization: Non-Hispanic White | 177 | 189 |  |  | 366
    Stage 1 Randomization: Non-Hispanic Black | 34 | 20 |  |  | 54
    Stage 1 Randomization: Hispanic, Any Race | 9 | 15 |  |  | 24
    Stage 1 Randomization: Other | 13 | 11 |  |  | 24
    Stage 2 Re-Randomization: number analyzed (Participants) | 0 | 0 | 132 | 127 | 259
    Stage 2 Re-Randomization: Non-Hispanic White |  |  | 103 | 96 | 199
    Stage 2 Re-Randomization: Non-Hispanic Black |  |  | 18 | 15 | 33
    Stage 2 Re-Randomization: Hispanic, Any Race |  |  | 4 | 8 | 12
    Stage 2 Re-Randomization: Other |  |  | 7 | 8 | 15
Weight [Mean (Standard Deviation); unit: pounds] — Population: We report data for two periods: "Stage 1 Randomization" (initial randomization to Week 3 or Week 7 Treatment Response Assessment) and "Stage 2 Re-Randomization" (re-randomization of sub-optimal responders to Portion controlled meals or Acceptance-based treatment).
  pounds
    Stage 1 Randomization: number analyzed (Participants) | 233 | 235 | 0 | 0 | 468
    Stage 1 Randomization | 225.1 (34.82) | 224.1 (34.25) |  |  | 224.6 (34.50)
    Stage 2 Re-Randomization: number analyzed (Participants) | 0 | 0 | 132 | 127 | 259
    Stage 2 Re-Randomization |  |  | 222.8 (34.55) | 222 (33.37) | 222.4 (33.91)

OUTCOME MEASURES:

1. Primary Outcome: Weight Change
Description: Weight change from baseline to 6 months and to 18 months among suboptimal responders to behavioral weight loss therapy.
Time Frame: 6 months and 18 months after baseline
Population: Participants included in this analysis were suboptimal responders to behavioral weight loss therapy whose initial treatment was augmented with portion-controlled meals or switched to acceptance-based treatment.
Measure: Mean (95% Confidence Interval); unit: pounds
Groups:
- Portion-controlled Meals: Portion-controlled meals: Participants continue with behavioral weight loss therapy, but this is augmented with portion-controlled meals (PCM).
- Acceptance-based Treatment: Acceptance-based treatment: Participants switch to treatment teaching acceptance-based behavioral skills.
Arm/Group | Portion-controlled Meals | Acceptance-based Treatment
Number analyzed (Participants) | 132 | 127
pounds
  6M | -18.4 [-20.5 to -16.2] | -15.7 [-18.0 to -13.4]
  18M | -8.5 [-10.7 to -6.3] | -7.4 [-9.7 to -5.2]
Statistical Analysis 1: Comparison: Portion-controlled Meals vs Acceptance-based Treatment; H1 predicted that suboptimal responders re-randomized to PCM would lose more weight at 6m (H1a) while those re-randomized to ABT would lose more weight at 18m (H1b). A mixed linear model predicted weight change from fixed re-randomization, measurement time, the re-randomization by measurement time interaction and covariate parameters; Test type: Superiority; p = 0.25, Mixed Models Analysis — 2 df re-random*time interaction tested if baseline to 6M or 18M PCM and ABT weight changes differed; primary hypothesis tests were 2 planned contrasts estimating baseline to 6M (H1a, expected neg) and 18M (H1b, expected pos) PCM vs. ABT weight change; The mixed model included a random participant intercept. Fixed covariates were baseline weight, TRA timing, sex, weight loss rate; The primary hypothesis tests were two planned contrasts that estimated weight change from baseline to 6M and 18M relative to baseline in PCM relative to ABT. A mixed linear model predicted weight changes between baseline and post-baseline for suboptimal responders, and this model included two a priori simple effects tests resulting in two mean differences, confidence intervals, and p-values. H1a: -2.7 lbs; 95% CI: -5.8, 0.5; p=0.09. H1b: -1.0 lbs; 95% CI: -4.2, 2.2; p=0.53

2. Secondary Outcome: Weight Change
Description: Mixed model-estimated weight change from baseline to 6 and 18 months (pooled) among all randomized participants.
Time Frame: 6 and 18 months after baseline
Population: Participants included in this analysis were all randomized participants, who had been randomly assigned to be assessed for treatment response 3 weeks (Early TRA) or 7 weeks (Late TRA) after initiating behavioral weight loss therapy.
Measure: Mean (95% Confidence Interval); unit: pounds
Groups:
- 3 Week Treatment Response Assessment (Early TRA): Participants all began by receiving Standard Behavioral Weight Loss Treatment (SBT) sessions. Participants were randomized to treatment response assessment (TRA) at Week 3.
- 7 Week Treatment Response Assessment (Late TRA): Participants all began by receiving Standard Behavioral Weight Loss Treatment (SBT) sessions. Participants were randomized to treatment response assessment (TRA) at Week 7.
Arm/Group | 3 Week Treatment Response Assessment (Early TRA) | 7 Week Treatment Response Assessment (Late TRA)
Number analyzed (Participants) | 233 | 235
pounds | -16.6 [-18.3 to -14.9] | -16.7 [-18.4 to -15.0]
Statistical Analysis 1: Comparison: 3 Week Treatment Response Assessment (Early TRA) vs 7 Week Treatment Response Assessment (Late TRA); Hypothesis 2 predicted that among all participants, those randomized to Early TRA would lose more weight at 6 and 18 months than those randomized to Late TRA. A mixed linear model predicted weight change from fixed treatment response assessment timing and covariate parameters; Test type: Superiority; p = 0.96, Mixed Models Analysis; The mixed model included a random participant intercept. Fixed covariates were baseline weight, sex, TRA result (PCM, ABT, responder, pre-TRA quit); Mean Difference (Net) = -0.1, 95% CI 2-sided [-2.4 to 2.3]

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Week 3 Treatment Response Assessment: Participants randomized to treatment response assessment at session 3. All participants start with standard behavioral weight loss treatment, and treatment response assessment occurs at session 3. If participants lost the expected amount of weight, no re-randomization occurs and participants continue with standard behavioral weight loss treatment. If participants did not lose the expected amount of weight, re-randomization to PCM or ABT occurs.
- Week 7 Treatment Response Assessment: Participants randomized to treatment response assessment at session 7. All participants start with standard behavioral weight loss treatment, and treatment response assessment occurs at session 7. If participants lost the expected amount of weight, no re-randomization occurs and participants continue with standard behavioral weight loss treatment. If participants did not lose the expected amount of weight, re-randomization to PCM or ABT occurs.
- Portion Controlled Meals: Portion controlled meals: Participants did not lose enough weight at the treatment response assessment (occurs at session 3 or session 7) and were re-randomized to portion controlled meals.
- Acceptance-based Treatment: Acceptance-based treatment: Participants did not lose enough weight at the treatment response assessment (occurs at session 3 or session 7) and were re-randomized to acceptance-based treatment.
Arm/Group | Week 3 Treatment Response Assessment | Week 7 Treatment Response Assessment | Portion Controlled Meals | Acceptance-based Treatment
All-Cause Mortality (participants affected / at risk) | 0/233 | 0/235 | 0/132 | 0/127
Serious Adverse Events (participants affected / at risk) | 0/233 | 3/235 | 1/132 | 2/127
Other Adverse Events (participants affected / at risk) | 0/233 | 0/235 | 0/132 | 0/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Week 3 Treatment Response Assessment (N=233) | Week 7 Treatment Response Assessment (N=235) | Portion Controlled Meals (N=132) | Acceptance-based Treatment (N=127)
Depressive disorders (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Kidney infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian cancer (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dehydration & Hypertension (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/02/NCT02368002/Prot_SAP_000.pdf